CLINICAL TRIAL: NCT02629965
Title: A Randomised, Double-blinded, Active-controlled 2-way Cross Over Trial to Assess the Effects of 6 Weeks Treatment of Once Daily Orally Inhaled Tiotropium + Olodaterol Fixed Dose Combination Delivered by RESPIMAT Inhaler Compared With Tiotropium Delivered by RESPIMAT Inhaler on Lung Hyperinflation, Exercise Capacity and Physical Activity in Japanese Patients With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Comparing the Efficacy of Tiotropium + Olodaterol Fixed Dose Combination (FDC) Over Tiotropium in Improvement of Lung Hyperinflation, Exercise Capacity and Physical Activity in Japanese COPD Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1237.33
Record Dates: First submitted 2015-12-01; First posted 2015-12-15 (Estimated); Results first posted 2019-06-06 (Actual); Last update posted 2019-06-06 (Actual); Status verified 2018-10

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide; olodaterol

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- tiotropium + olodaterol (Experimental): inhalation two puffs from the RESPIMAT inhaler, once a day, in the morning
  Interventions: Drug: tiotropium; Drug: olodaterol
- tiotropium (Active Comparator): inhalation two puffs from the RESPIMAT inhaler, once a day, in the morning
  Interventions: Drug: tiotropium

INTERVENTIONS:
Drug: tiotropium — fixed dose combination
  Arms: tiotropium + olodaterol
Drug: olodaterol — fixed dose combination
  Arms: tiotropium + olodaterol
Drug: tiotropium
  Arms: tiotropium

SUMMARY:
This is a multi-centre, randomised, double-blinded, active-controlled, 2-way cross over trial to assess the effects of once daily administration of orally inhaled tiotropium + olodaterol FDC or tiotropium (both delivered by the RESPIMAT Inhaler) on pulmonary function (lung hyperinflation), exercise capacity (6-minute walk distance) and physical activities after 6 weeks of treatment in Japanese patients with Chronic Obstructive Pulmonary Disease.

ELIGIBILITY:
Inclusion criteria:

* All patients must sign an informed consent consistent with International Conference on Harmonization - Good Clinical Practice (ICH-GCP) guidelines prior to participation in the trial, which includes medication washout and restrictions.
* All patients must have a diagnosis of chronic obstructive pulmonary disease (COPD) and must meet the following spirometric criteria:

Patients must have relatively stable airway obstruction with a post-bronchodilator Forced expiratory volume in one second (FEV1) < 80% of predicted normal and post-bronchodilator FEV1/forced vital capacity (FVC) < 70% at Visit 1.

* Male or female patients, aged >= 40 years.
* Patients must be current or ex-smokers with a smoking history of more than 10 pack years. Patients who have never smoked cigarettes must be excluded.
* Patients with score on the modified Medical Research Council (mMRC) >= 1.
* Patients who walk < 400 meters of 6MWT and have a score on the modified Borg >= 4 at the end of 6 minute walk test (6MWT) at Visit 2.
* Patients must be able to perform technically acceptable pulmonary function tests (spirometry), to use the physical activity monitor and must be able to complete 6MWT during the study period as required in the protocol.
* Patients must be able to inhale medication in a competent manner from the RESPIMAT Inhaler and from a metered dose inhaler.

Exclusion criteria:

* Patients with a significant disease other than COPD; a significant disease is defined as a disease which, in the opinion of the investigator, may put the patient at risk because of participation in the study, influence the results of the study and cause concern regarding the patient's ability to participate in the study.
* Patients with clinically relevant abnormal baseline haematology, blood chemistry,urinalysis or creatinine > x2 upper limit of normal (ULN) will be excluded regardless of clinical condition (a repeat laboratory evaluation can be conducted if deemed necessary by the investigator).
* Patients with a current documented diagnosis of asthma. For patients with allergic rhinitis or atopy, source documentation is required to verify that the patient does not have asthma.
* Further exclusion criteria apply

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2016-02-12 (Actual); Primary Completion 2017-03-24 (Actual); Study Completion 2017-04-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (43):
- Japan (43):
  - Hiramatsu Internal and Respiratory Medicine Clinic, Aichi, Komaki
  - National Hospital for Geriatric Medicine, Aichi, Obu
  - Tosei General Hospital, Aichi, Seto
  - Nishi Fukuoka Hospital, Fukuoka, Fukuoka
  - Kirigaoka Tsuda Hospital, Fukuoka, Kitakyushu
  - Osaki Internal and Respiratory Clinic, Fukuoka, Kitakyushu
  - Kurume University Hospital, Fukuoka, Kurume
  - Tohno Chuo Clinic, Gifu, Mizunami
  - Mazda Hospital, Hiroshima, Aki-gun
  - Teine Keijinkai Clinic, Hokkaido, Sapporo
  - Hokkaido University Hospital, Hokkaido, Sapporo
  - KKR Sapporo Medical Center, Hokkaido, Sapporo
  - Japan Community Health Care Organization Hokkaido Hospital, Hokkaido, Sapporo
  - Kobe City Medical Center General Hospital, Hyogo, Kobe
  - Kobe City Hospital Organization Kobe City Medical Center West Hospital, Hyogo, Kobe
  - Ibarakihigashi National Hospial, Ibaraki, Naka-gun
  - Iwate Medical University Hospital, Iwate, Morioka
  - Sakaide City Hospital, Kagawa, Sakaide
  - Kagoshima University Medical And Dental Hospital, Kagoshima, Kagoshima
  - Kokan Clinic, Kanagawa, Kawasaki
  - Shin-yurigaoka General Hospital, Kanagawa, Kawasaki
  - Showa University Fujigaoka Hospital, Kanagawa, Yokohama
  - Kyoto University Hospital, Kyoto, Kyoto
  - Rakuwakai Otowa Hospital, Kyoto, Kyoto
  - Uji-Tokushukai Medical Center, Kyoto, Uji
  - Matsusaka City Hospital, Mie, Matsusaka
  - Tohoku University Hospital, Miyagi, Sendai
  - Tohoku Rosai Hospital, Miyagi, Sendai
  - Kishiwada City Hospital, Osaka, Kishiwada
  - Kindai University Hospital, Osaka, Osakasayama
  - Osaka City University Hospital, Osaka, Osaka
  - National Hospital Organization Toneyama National Hospital, Osaka, Toyonaka
  - Yao Tokushukai General Hospital, Osaka, Yao
  - Shimane University Hospital, Shimane, Izumo
  - Tenryu Hospital, Shizuoka, Hamamatsu
  - Juntendo University Hospital, Tokyo, Bunkyo-ku
  - The Respiratory Care Clinic, Nippon Medical School, Tokyo, Chiyoda-ku
  - Nihonbashi Sakura Clinic, Tokyo, Chuo-ku
  - Tokyo Medical University Hachioji Medical Center, Tokyo, Hachioji
  - Nihon University Itabashi Hospital, Tokyo, Itabashi-ku
  - Showa University Hospital, Tokyo, Shinagawa-ku
  - Shinjuku Research Park Clinic, Tokyo, Shinjuku-ku
  - Wakayama National Hospital, Wakayama, Hidaka-gun

REFERENCES:
- [Derived] Minakata Y, Motegi T, Ueki J, Gon Y, Nakamura S, Anzai T, Hirata K, Ichinose M. Effect of tiotropium/olodaterol on sedentary and active time in patients with COPD: post hoc analysis of the VESUTO(R) study. Int J Chron Obstruct Pulmon Dis. 2019 Aug 7;14:1789-1801. doi: 10.2147/COPD.S208081. eCollection 2019. PMID 31496678

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a randomised, double-blind, active-controlled, 2-way crossover trial to assess the effects of once daily treatment of orally inhaled Tiotropium + Olodaterol FDC 5 μg/5 μg or Tiotropium 5 μg over 12 weeks of treatment in Japanese patients with Chronic obstructive pulmonary disease (COPD).
Pre-assignment Details: All patients were screened for eligibility to participate in the trial. Subjects attended specialist sites which would then ensure that all subjects met all inclusion/exclusion criteria. Subjects were not to be randomised to trial treatment if any one of the specific entry criteria were violated.
Groups:
- Tiotropium 5 μg / Tiotropium + Olodaterol 5/5 μg FDC: Participants inhaled 2 puffs from the RESPIMAT Inhaler of the Tiotropium inhalation solution (2.5 microgram per actuation) in period 1 and Tiotropium + Olodaterol inhalation solution (2.5/2.5 microgram per actuation) in period 2 once a day in the morning for a total of 12 weeks
  2 treatments were not separated by wash-out periods.
- Tiotropium + Olodaterol 5/5 μg FDC / Tiotropium 5 μg: Participants inhaled 2 puffs from the RESPIMAT Inhaler of the Tiotropium + Olodaterol inhalation solution (2.5/2.5 microgram per actuation) in period 1 and Tiotropium inhalation solution (2.5 microgram per actuation) in period 2 once a day in the morning for a total of 12 weeks.
  2 treatments were not separated by wash-out periods.
Period: Period 1
Arm/Group | Tiotropium 5 μg / Tiotropium + Olodaterol 5/5 μg FDC | Tiotropium + Olodaterol 5/5 μg FDC / Tiotropium 5 μg
Started | 92 | 92
Completed | 88 | 90
Not Completed | 4 | 2
Not completed — Adverse Event | 1 | 0
Not completed — Unexpected worsening of disease | 2 | 0
Not completed — Other than listed above | 1 | 2
Period: Period 2
Arm/Group | Tiotropium 5 μg / Tiotropium + Olodaterol 5/5 μg FDC | Tiotropium + Olodaterol 5/5 μg FDC / Tiotropium 5 μg
Started | 88 | 90
Completed | 87 | 90
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): Treated set includes all particiapatns who took at least one study medication.
Groups:
- Total: Total randomised participants in the trial.
Arm/Group | Total
Number analyzed (Participants) | 184
Age, Continuous [Mean (Standard Deviation); unit: Years] — The age data are presented by years. Population: Treated set (TS): TS includes patients who had baseline measurement and at least 1 post-baseline measurement for the primary endpoint or a secondary endpoint.
  Years | 72.8 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants] — The sex data are presented by count of participants. Population: Treated set (TS): TS includes patients who had baseline measurement and at least 1 post-baseline measurement for the primary endpoint or a secondary endpoint.
  Participants
    Female | 19
    Male | 165
Race (NIH/OMB) [Count of Participants; unit: Participants] — The race data are presented by count of participants. Ethnicity was not collected for this study. Population: Treated set (TS): TS includes patients who had baseline measurement and at least 1 post-baseline measurement for the primary endpoint or a secondary endpoint.
  Participants
    American Indian or Alaska Native | 0
    Asian | 184
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 0
    White | 0
    More than one race | 0
    Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Inspiratory Capacity at Rest Measured at 60 Minutes Post-dose
Description: At day 43 inspiratory capacity at rest measured at 60 minutes post-dose, after 6 weeks of each treatment. Adjusted mean was entered instead of mean in statistical analysis.
Time Frame: Day 43, 60 minutes post-dose after 6 weeks of each treatment
Population: Full analysis set (FAS): FAS includes participants who had baseline measurement and at least 1 post-baseline measurement for the primary endpoint or a secondary endpoint. The FAS was used for the efficacy analyses.
Measure: Mean (Standard Error); unit: Litre (L)
Groups:
- Tiotropium 5 μg: Participants inhaled 2 puffs from the RESPIMAT Inhaler of the Tiotropium inhalation solution (2.5 microgram per actuation) once a day in the morning for 2 periods for 6 weeks.
- Tiotropium + Olodaterol 5/5 μg: Participants inhaled 2 puffs from the RESPIMAT Inhaler of the Tiotropium + Olodaterol inhalation solution (2.5/2.5 microgram per actuation) once a day in the morning for 2 periods for 6 weeks.
Arm/Group | Tiotropium 5 μg | Tiotropium + Olodaterol 5/5 μg
Number analyzed (Participants) | 178 | 179
Litre (L) | 1.875 (0.019) | 1.990 (0.019)
Statistical Analysis 1: Comparison: Tiotropium 5 μg vs Tiotropium + Olodaterol 5/5 μg; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mixed Effect Model Repeated Measures includes treatment and period as fixed effects, study baseline as a covariate and patient as a random effect; Mean Difference (Final Values) = 0.115, 95% CI 2-sided [0.077 to 0.153], Standard Error of Mean 0.019 — Adjusted mean of differences between treatments and standard error; Mixed effect repeated measurement was used to calculate adjusted mean values as well as treatment contrasts together with the 95% confidence intervals (CIs) and p-values

2. Secondary Outcome: 6-minute Walk Distance [Meter]
Description: 6-minute walk distance [Meter] treatment comparisons after 6 weeks of each treatment. Adjusted mean was entered instead of mean in statistical analysis.
Time Frame: Day 43, 60 minutes post-dose after 6 weeks of each treatment
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Meter (m)
Arm/Group | Tiotropium 5 μg | Tiotropium + Olodaterol 5/5 μg
Number analyzed (Participants) | 178 | 178
Meter (m) | 307.356 (5.170) | 311.524 (5.170)
Statistical Analysis 1: Comparison: Tiotropium 5 μg vs Tiotropium + Olodaterol 5/5 μg; Test type: Superiority; p = 0.4291, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 4.168, 95% CI 2-sided [-6.211 to 14.548], Standard Error of Mean 5.260 — Adjusted mean of differences between treatments and standard error; [other analysis details as in outcome 1, analysis 1]

3. Secondary Outcome: Average Number of Step Per Day (Step/Day)
Description: At day 43 adjusted mean (SE) of average number of step per day [step/day] treatment comparisons in measured by the activity monitor in 2 weeks prior to Week 6 of each treatment. Adjusted mean was entered instead of mean in statistical analysis.
Time Frame: 2 weeks prior to Week 6 per treatment
Population: as for outcome 1
Measure: Mean (Standard Error); unit: step/day
Arm/Group | Tiotropium 5 μg | Tiotropium + Olodaterol 5/5 μg
Number analyzed (Participants) | 179 | 179
step/day | 3550.400 (93.123) | 3559.901 (93.460)
Statistical Analysis 1: Comparison: Tiotropium 5 μg vs Tiotropium + Olodaterol 5/5 μg; Test type: Superiority; p = 0.9098, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 9.501, 95% CI 2-sided [-155.692 to 174.694], Standard Error of Mean 83.704 — Adjusted mean of differences between treatments and standard error; [other analysis details as in outcome 1, analysis 1]

4. Secondary Outcome: Average Daily Duration (Minutes) of ≥ 4 Metabolic Equivalents (METs)
Description: At day 43 adjusted mean (SE) of average daily duration [minute] of ≥ 4 METs treatment comparisons measured by the activity monitor in the 2 weeks prior to week 6 of each treatment. Adjusted mean was entered instead of mean in statistical analysis.
Time Frame: 2 weeks prior to Week 6 per treatment
Population: as for outcome 1
Measure: Mean (Standard Error); unit: minute
Arm/Group | Tiotropium 5 μg | Tiotropium + Olodaterol 5/5 μg
Number analyzed (Participants) | 179 | 177
minute | 10.206 (0.497) | 9.914 (0.499)
Statistical Analysis 1: Comparison: Tiotropium 5 μg vs Tiotropium + Olodaterol 5/5 μg; Test type: Superiority; p = 0.5338, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.292, 95% CI 2-sided [-1.217 to 0.633], Standard Error of Mean 0.469 — Adjusted mean of differences between treatments and standard error; [other analysis details as in outcome 1, analysis 1]

5. Secondary Outcome: Average Daily Duration (Minutes) of ≥ 3 Metabolic Equivalents (METs)
Description: At day 43 adjusted mean (SE) of average daily duration [minute] of ≥ 3 METs treatment comparisons measured by the activity monitor in 2 weeks prior to Week 6 of each treatment. Adjusted mean was entered instead of mean in statistical analysis.
Time Frame: 2 weeks prior to Week 6 per treatment
Population: as for outcome 1
Measure: Mean (Standard Error); unit: minute
Arm/Group | Tiotropium 5 μg | Tiotropium + Olodaterol 5/5 μg
Number analyzed (Participants) | 179 | 177
minute | 44.662 (0.979) | 45.601 (0.979)
Statistical Analysis 1: Comparison: Tiotropium 5 μg vs Tiotropium + Olodaterol 5/5 μg; Test type: Superiority; p = 0.3524, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.939, 95% CI 2-sided [-1.048 to 2.926], Standard Error of Mean 1.007 — Adjusted mean of differences between treatments and standard error; [other analysis details as in outcome 1, analysis 1]

6. Secondary Outcome: Average Daily Duration (Minutes) of ≥ 2 Metabolic Equivalents (METs)
Description: At day 43 adjusted mean (SE) of average daily duration [minute] of ≥ 2 METs treatment comparison measured by the activity monitor in 2 weeks prior to Week 6 of each treatment. Adjusted mean was entered instead of mean in statistical analysis.
Time Frame: 2 weeks prior to Week 6 per treatment
Population: as for outcome 1
Measure: Mean (Standard Error); unit: minute
Arm/Group | Tiotropium 5 μg | Tiotropium + Olodaterol 5/5 μg
Number analyzed (Participants) | 179 | 177
minute | 171.935 (2.506) | 174.192 (2.517)
Statistical Analysis 1: Comparison: Tiotropium 5 μg vs Tiotropium + Olodaterol 5/5 μg; Test type: Superiority; p = 0.3949, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 2.257, 95% CI 2-sided [-2.966 to 7.481], Standard Error of Mean 2.647 — Adjusted mean of differences between treatments and standard error; [other analysis details as in outcome 1, analysis 1]

7. Secondary Outcome: Average Daily Active Strength (Metabolic Equivalents*Minutes) of ≥ 3 METs
Description: At day 43 adjusted mean (SE) of average daily active strength [METs x minute] of >=3 METs treatment comparisons measured by the activity monitor in 2 weeks prior to Week 6 of each treatment. Adjusted mean was entered instead of mean in statistical analysis.
Time Frame: 2 weeks prior to Week 6 per treatment
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Metabolic equivalents * minutes
Arm/Group | Tiotropium 5 μg | Tiotropium + Olodaterol 5/5 μg
Number analyzed (Participants) | 179 | 177
Metabolic equivalents * minutes | 148.647 (3.723) | 151.067 (3.737)
Statistical Analysis 1: Comparison: Tiotropium 5 μg vs Tiotropium + Olodaterol 5/5 μg; Test type: Superiority; p = 0.4955, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 2.420, 95% CI 2-sided [-4.572 to 9.411], Standard Error of Mean 3.543 — Adjusted mean of differences between treatments and standard error; [other analysis details as in outcome 1, analysis 1]

8. Secondary Outcome: 60 Minutes Post-dose Slow Vital Capacity (SVC) (in Litre)
Description: At day 43 adjusted mean (SE) of 60 minute post-dose slow vital capacity [Litre] treatment comparisons after 6 weeks of each treatment. Adjusted mean was entered instead of mean in statistical analysis.
Time Frame: Day 43, 60 minutes post-dose after 6 weeks of each treatment
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Litre (L)
Arm/Group | Tiotropium 5 μg | Tiotropium + Olodaterol 5/5 μg
Number analyzed (Participants) | 178 | 179
Litre (L) | 2.962 (0.021) | 3.096 (0.021)
Statistical Analysis 1: Comparison: Tiotropium 5 μg vs Tiotropium + Olodaterol 5/5 μg; Test type: Superiority; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.134, 95% CI 2-sided [0.091 to 0.176], Standard Error of Mean 0.022 — Adjusted mean of differences between treatments and standard error; [other analysis details as in outcome 1, analysis 1]

9. Secondary Outcome: 30 Minutes Post-dose Forced Expiratory Volume in One Second (FEV1) (in Litre)
Description: At day 43 adjusted mean (SE) of 30 minute post-dose forced expiratory volume in one second (FEV1) [Litre] treatment comparisons after 6 weeks of each treatment. Adjusted mean was entered instead of mean in statistical analysis.
Time Frame: Day 43, 30 minutes post-dose after 6 weeks of each treatment
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Litre (L)
Arm/Group | Tiotropium 5 μg | Tiotropium + Olodaterol 5/5 μg
Number analyzed (Participants) | 180 | 179
Litre (L) | 1.169 (0.011) | 1.275 (0.011)
Statistical Analysis 1: Comparison: Tiotropium 5 μg vs Tiotropium + Olodaterol 5/5 μg; Test type: Superiority; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.105, 95% CI 2-sided [0.088 to 0.123], Standard Error of Mean 0.009 — Adjusted mean of differences between treatments and standard error; [other analysis details as in outcome 1, analysis 1]

10. Secondary Outcome: 30 Minutes Post-dose Forced Vital Capacity (FVC) (in Litre)
Description: At day 43 adjusted mean (SE) of 30 minute post-dose forced vital capacity (FVC) [Litre] treatment comparisons after 6 weeks of each treatment. Adjusted mean was entered instead of mean in statistical analysis.
Time Frame: Day 43, 30 minutes post-dose after 6 weeks of each treatment
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Litre (L)
Arm/Group | Tiotropium 5 μg | Tiotropium + Olodaterol 5/5 μg
Number analyzed (Participants) | 180 | 179
Litre (L) | 2.857 (0.021) | 3.020 (0.021)
Statistical Analysis 1: Comparison: Tiotropium 5 μg vs Tiotropium + Olodaterol 5/5 μg; Test type: Superiority; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.163, 95% CI 2-sided [0.130 to 0.197], Standard Error of Mean 0.017 — Adjusted mean of differences between treatments and standard error; [other analysis details as in outcome 1, analysis 1]

11. Post Hoc Outcome: Inspiratory Capacity [Litre] Treatment Comparisons of 6-Minute Walk Test (6MWT) Completer at Treatment Period
Description: At day 43 adjusted mean (standard error) of inspiratory capacity [Litre] test comparisons after 6 weeks of each treatment for 6MWT completer at treatment period. Adjusted mean was entered instead of mean in statistical analysis.
Time Frame: Day 43, 60 minutes post-dose after 6 weeks of each treatment
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Litre (L)
Arm/Group | Tiotropium 5 μg | Tiotropium + Olodaterol 5/5 μg
Number analyzed (Participants) | 119 | 121
Litre (L) | 1.940 (0.022) | 2.072 (0.022)
Statistical Analysis 1: Comparison: Tiotropium 5 μg vs Tiotropium + Olodaterol 5/5 μg; Test type: Superiority; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.133, 95% CI 2-sided [0.103 to 0.162], Standard Error of Mean 0.015 — Adjusted mean of differences between treatments and standard error; [other analysis details as in outcome 1, analysis 1]

12. Post Hoc Outcome: Inspiratory Capacity [Litre] Treatment Comparisons of 6-Minute Walk Test (6MWT) Completer at Baseline Period
Description: At day 43 adjusted mean (standard error) of inspiratory capacity [Litre] test comparisons after 6 weeks of each treatment for 6MWT completer at baseline period. Adjusted mean was entered instead of mean in statistical analysis.
Time Frame: Day 43, 60 minutes post-dose after 6 weeks of each treatment
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Litre (L)
Arm/Group | Tiotropium 5 μg | Tiotropium + Olodaterol 5/5 μg
Number analyzed (Participants) | 128 | 128
Litre (L) | 1.925 (0.021) | 2.053 (0.021)
Statistical Analysis 1: Comparison: Tiotropium 5 μg vs Tiotropium + Olodaterol 5/5 μg; Test type: Superiority; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.128, 95% CI 2-sided [0.100 to 0.156], Standard Error of Mean 0.014 — Adjusted mean of differences between treatments and standard error; [other analysis details as in outcome 1, analysis 1]

13. Post Hoc Outcome: Inspiratory Capacity [Litre] Test Comparisons of 6-Minute Walk Treatment (6MWT) in-Completer at Treatment Period
Description: At day 43 adjusted mean (standard error) of inspiratory capacity [Litre] test comparisons after 6 weeks of each treatment for 6MWT in-completer at treatment period. Adjusted mean was entered instead of mean in statistical analysis.
Time Frame: Day 43, 60 minutes post-dose after 6 weeks of each treatment
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Litre (L)
Arm/Group | Tiotropium 5 μg | Tiotropium + Olodaterol 5/5 μg
Number analyzed (Participants) | 59 | 58
Litre (L) | 1.738 (0.024) | 1.820 (0.024)
Statistical Analysis 1: Comparison: Tiotropium 5 μg vs Tiotropium + Olodaterol 5/5 μg; Test type: Superiority; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.082, 95% CI 2-sided [0.056 to 0.108], Standard Error of Mean 0.013 — Adjusted mean of differences between treatments and standard error; [other analysis details as in outcome 1, analysis 1]

14. Post Hoc Outcome: Inspiratory Capacity [Litre] Treatment Comparisons of 6-Minute Walk Test (6MWT) in-Completer at Baseline Period
Description: At day 43 adjusted mean (standard error) of inspiratory capacity [Litre] test comparisons after 6 weeks of each test for 6MWT in-completer at baseline period. Adjusted mean was entered instead of mean in statistical analysis.
Time Frame: Day 43, 60 minutes post-dose after 6 weeks of each treatment
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Litre (L)
Arm/Group | Tiotropium 5 μg | Tiotropium + Olodaterol 5/5 μg
Number analyzed (Participants) | 50 | 51
Litre (L) | 1.744 (0.026) | 1.830 (0.026)
Statistical Analysis 1: Comparison: Tiotropium 5 μg vs Tiotropium + Olodaterol 5/5 μg; Test type: Superiority; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.086, 95% CI 2-sided [0.058 to 0.114], Standard Error of Mean 0.014 — Adjusted mean of differences between treatments and standard error; [other analysis details as in outcome 1, analysis 1]

15. Post Hoc Outcome: Inspiratory Capacity [Litre] Treatment Comparisons of Subgroup of Global Initiative for Chronic Obstructive Lung Disease (GOLD) Stage I/II
Description: At day 43 adjusted mean (standard error) of inspiratory capacity [Litre] treatment comparisons after 6 weeks of each treatment for subgroup of GOLD stage I/II. Adjusted mean was entered instead of mean in statistical analysis.
Time Frame: Day 43, 60 minutes post-dose after 6 weeks of each treatment
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Litre (L)
Arm/Group | Tiotropium 5 μg | Tiotropium + Olodaterol 5/5 μg
Number analyzed (Participants) | 97 | 97
Litre (L) | 2.023 (0.023) | 2.106 (0.023)
Statistical Analysis 1: Comparison: Tiotropium 5 μg vs Tiotropium + Olodaterol 5/5 μg; Test type: Superiority; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.083, 95% CI 2-sided [0.059 to 0.108], Standard Error of Mean 0.012 — Adjusted mean of differences between treatments and standard error; [other analysis details as in outcome 1, analysis 1]

16. Post Hoc Outcome: Inspiratory Capacity [Litre] Treatment Comparisons of Subgroup of Global Initiative for Chronic Obstructive Lung Disease (GOLD) Stage III/IV
Description: At day 43 adjusted mean (standard error) of inspiratory capacity [Litre] treatment comparisons after 6 weeks of each treatment for subgroup of GOLD stage III/IV. Adjusted mean was entered instead of mean in statistical analysis.
Time Frame: Day 43, 60 minutes post-dose after 6 weeks of each treatment
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Litre (L)
Arm/Group | Tiotropium 5 μg | Tiotropium + Olodaterol 5/5 μg
Number analyzed (Participants) | 81 | 82
Litre (L) | 1.697 (0.026) | 1.849 (0.026)
Statistical Analysis 1: Comparison: Tiotropium 5 μg vs Tiotropium + Olodaterol 5/5 μg; Test type: Superiority; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.152, 95% CI 2-sided [0.114 to 0.189], Standard Error of Mean 0.019 — Adjusted mean of differences between treatments and standard error; [other analysis details as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: From first drug administration until 12 weeks after last drug administration, up to 15 weeks
Description: An adverse event was defined as any untoward medical occurrence in a patient or clinical investigation participants administered a trial medicine.
Groups:
- Tiotropium 5: Participants were orally inhaled 2 puffs from the RESPIMAT Inhaler with the Tiotropium fixed dose combination of 2.5 μg per actuation once a day in the morning for 6 weeks.
- Tiotropium + Olodaterol 5/5: Participants were orally inhaled 2 puffs from the RESPIMAT Inhaler with the Tiotropium + Olodaterol fixed dose combination of 2.5/2.5 μg per actuation once a day in the morning for 6 weeks.
Arm/Group | Tiotropium 5 | Tiotropium + Olodaterol 5/5
All-Cause Mortality (participants affected / at risk) | 0/182 | 0/180
Serious Adverse Events (participants affected / at risk) | 7/182 | 7/180
Other Adverse Events (participants affected / at risk) | 11/182 | 18/180
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tiotropium 5 (N=182) | Tiotropium + Olodaterol 5/5 (N=180)
Vertigo positional (Ear and labyrinth disorders) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Vestibular neuronitis (Infections and infestations) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Bladder cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Altered state of consciousness (Nervous system disorders) | 0 | 1
Renal impairment (Renal and urinary disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Aortic aneurysm (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tiotropium 5 (N=182) | Tiotropium + Olodaterol 5/5 (N=180)
Viral upper respiratory tract infection (Infections and infestations) | 11 | 18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-04-10): https://cdn.clinicaltrials.gov/large-docs/65/NCT02629965/SAP_000.pdf
  • Study Protocol (2015-10-30): https://cdn.clinicaltrials.gov/large-docs/65/NCT02629965/Prot_001.pdf